CLINICAL TRIAL: NCT01097096
Title: A 90-week, Multi-center, Randomized, Double-blind, Placebo-controlled Study in Patients With Mild Alzheimer's Disease (AD) to Investigate the Safety, Tolerability and Abeta-specific Antibody Response Following Repeated i.m. Injections of Adjuvanted CAD106
Brief Title: Safety, Tolerability and Abeta-specific Antibody Response of Repeated i.m. Injections of Adjuvanted CAD106 in Mild Alzheimer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCAD106A2203; 2009-012394-35 (EudraCT Number)
Record Dates: First submitted 2010-03-29; First posted 2010-04-01 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Alzheimer's Disease
Keywords: Active immunization; Alzheimer disease; Antibody; Central Nervous System Diseases; Neurodegenerative diseases; Vaccine
MeSH Terms: conditions — Alzheimer Disease; Central Nervous System Diseases; Neurodegenerative Diseases | interventions — aluminum sulfate; MF59 oil emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (9):
- CAD106 150μg + Adjuvant 1 at middle dose (Active Comparator)
  Interventions: Biological: CAD106; Biological: MF59
- CAD106 150μg + Adjuvant 1 at low dose (Active Comparator)
  Interventions: Biological: CAD106; Biological: MF59
- Placebo + Adjuvant 1 at middle dose (Placebo Comparator)
  Interventions: Biological: Placebo
- CAD106 150μg + Adjuvant 2 at middle dose (Active Comparator)
  Interventions: Biological: CAD106; Biological: MF59
- CAD106 150μg + Adjuvant 2 at low dose (Active Comparator)
  Interventions: Biological: CAD106; Biological: MF59
- Placebo + Adjuvant 2 at middle dose (Placebo Comparator)
  Interventions: Biological: Placebo
- CAD106 450μg + either Adjuvant 1 or 2 at middle dose (Active Comparator)
  Interventions: Biological: CAD106; Biological: Alum; Biological: MF59
- CAD106 450μg + either Adjuvant 1 or 2 at low dose (Active Comparator)
  Interventions: Biological: CAD106; Biological: Alum; Biological: MF59
- Placebo + either Adjuvant 1 or 2 at middle dose (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CAD106 — 150μg and 450μg doses were reconstituted and administered via intramuscular injection
  Arms: CAD106 150μg + Adjuvant 1 at low dose; CAD106 150μg + Adjuvant 1 at middle dose; CAD106 150μg + Adjuvant 2 at low dose; CAD106 150μg + Adjuvant 2 at middle dose; CAD106 450μg + either Adjuvant 1 or 2 at low dose; CAD106 450μg + either Adjuvant 1 or 2 at middle dose
Biological: Placebo — Identical placebo to CAD106 administered via intramuscular injection
  Arms: Placebo + Adjuvant 1 at middle dose; Placebo + Adjuvant 2 at middle dose; Placebo + either Adjuvant 1 or 2 at middle dose
Biological: Alum — An adjuvant (additive to increase potency ) of low, middle or high doses which was mixed with reconstituted active CAD106
  Arms: CAD106 450μg + either Adjuvant 1 or 2 at low dose; CAD106 450μg + either Adjuvant 1 or 2 at middle dose
Biological: MF59 — An adjuvant (additive to increase potency) of low, middle and high doses which was mixed with reconstituted active CAD106
  Arms: CAD106 150μg + Adjuvant 1 at low dose; CAD106 150μg + Adjuvant 1 at middle dose; CAD106 150μg + Adjuvant 2 at low dose; CAD106 150μg + Adjuvant 2 at middle dose; CAD106 450μg + either Adjuvant 1 or 2 at low dose; CAD106 450μg + either Adjuvant 1 or 2 at middle dose

SUMMARY:
This study will assess the safety, tolerability and Abeta-specific antibody response of repeated intra-muscular injections of adjuvanted CAD106 in patients with mild Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female patients below 85 years of age (inclusive)
* Diagnosis of mild Alzheimer's Disease
* Mini-Mental State Examination (MMSE) 20 to 26 (inclusive) at screening, untreated or on stable dose of cholinesterase inhibitor or memantine over the last 4 weeks prior to clinical assessments

Exclusion Criteria:

* Previously participated in an AD vaccine study and received active treatment
* History or presence of an active autoimmune disease
* History or presence of seizure disorder
* Presence of significant coronary heart disease and/or cerebrovascular disease
* Presence of other neurodegenerative disease and/or psychiatric disorders (with the exception of successfully treated depression)
* Advanced, severe, progressive or unstable disease that might interfere with the safety, tolerability and pharmacodynamic assessments of the patient

Other protocol-defined inclusion/exclusion criteria may apply

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessments (physical/neurological examinations, electrocardiogram (ECG), vital signs, standard and special laboratory evaluations, Magnetic Resonance Imaging (MRIs), Adverse events / Serious adverse events (AE/SAE) monitoring). | Screening and through the end of the study to Week 90

SECONDARY OUTCOMES:
Amyloid beta (Aβ)-specific and Qβ carrier-specific antibody response to CAD106 (with either adjuvant) in serum and cerebrospinal fluid (CSF) | Screening and through the end of the study to Week 90
Amyloid beta (Aβ)-specific and Qβ carrier-specific T-cell response to CAD106 (with either adjuvant) using peripheral blood mononuclear cells (PBMCs) | Screening and at week 8
Changes over time of the concentrations of disease related markers (Aβ1-40 and Aβ1-42 in plasma; Aβ1-40, Aβ1-42, total-tau, phospho-tau in CSF, or other markers) in patients with mild AD receiving CAD106 (with either adjuvant) compared to placebo | Screening and through the end of the study to Week 90

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- United States (5):
  - Novartis Investigative Site, Costa Mesa, California
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Eatontown, New Jersey
- Belgium (2):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Leuven
- Canada (3):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- Germany (2):
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Nuremberg
- Italy (5):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Stavanger, Norway
- Spain (3):
  - Novartis Investigative Site, Sant Cugat del Vallès, Barcelona
  - Novartis Investigative Site, Barakaldo, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
- Sweden (2):
  - Novartis Investigative Site, Mölndal
  - Novartis Investigative Site, Stockholm
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Biel
  - Novartis Investigative Site, Lausanne

REFERENCES:
- See also: Resuls for CCAD106A2203 on the Novartis Clinical Trial website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10603